CLINICAL TRIAL: NCT04992806
Title: A Retrospective Study on the Effect of Arthroscopy on Hip Diseases
Brief Title: A Retrospective Study on the Effect of Surgery on Hip Diseases
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-2016015
Record Dates: First submitted 2021-06-27; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-06

CONDITIONS: Femoroacetabular Impingement; Acetabular Labral Tear
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients accepted hip arthroscopy: patients with hip diseases and accepted hip arthroscopy in Peking University Third Hospital
  Interventions: Procedure: hip arthroscopy

INTERVENTIONS:
Procedure: hip arthroscopy — Use epidural anesthesia or general anesthesia. The patient lies on the orthopedic traction bed to protect the perineum and perform traction of the lower limbs on the surgical side. Under arthroscopy, check the labrum, acetabular articular surface and femoral head cartilage, and round ligament in turn. The acetabular labrum with tear degeneration was treated with labrum suture or labrum revision surgery according to the injury. Perform femoral head and neck plastic or acetabular plastic surgery, osteoid osteoma debridement, etc.

SUMMARY:
To study the effect of arthroscopy on the treatment of hip diseases and to evaluate the regularity and treatment of hip joint diseases.

DETAILED DESCRIPTION:
To study the clinical effect of arthroscopic treatment in patients with hip disease, a retrospective study was conducted on 600 patients with hip disease from January 2011 to January 2016. All patients underwent preoperative examinations. These included preoperative supine anteroposterior hip radiographs, cross-lateral radiographs, computed tomography (CT), and magnetic resonance imaging.Preoperative patient-reported outcomes (PROs), including visual analogue scale (VAS), international hip prognostic instrument-12 (IHOT-12), and modified Harris hip score (MHHS), were evaluated at 1, 2, and 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patient received imaging examination before surgery and was diagnosed with hip joint labrum injury, FAI and other hip joint diseases, and the patient complained of pain in the hip joint, buttocks or thigh. Conservative treatment is ineffective for more than 6 months.

Exclusion Criteria:

* History of hip surgery, hip osteoarthritis, femoral head necrosis, hip infection, rheumatic disease, lumbar disease, ankylosing spondylitis, or sacroiliac joint disease.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We evaluated consecutive patients who were diagnosed with hip diseases (i.e. FAI, Acetabulum labrum tear) and who underwent hip arthroscopy at our hospital between January 2011 and January 2016.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
The patient was followed up at 1 year after surgery to evaluate the Visual Analog Scale (VAS). | 1 year after operation
  Visual Analog Scale (VAS), The highest score was 10, and the lowest was 0. The higher the score, the more obvious the pain.
The patient was followed up at 2 years after surgery to evaluate the Visual Analog Scale (VAS). | 2 years after operation
  Visual Analog Scale (VAS), The highest score was 10, and the lowest was 0. The higher the score, the more obvious the pain.
The patient was followed up at 5 years after surgery to evaluate the Visual Analog Scale (VAS). | 5 years after operation
  Visual Analog Scale (VAS), The highest score was 10, and the lowest was 0. The higher the score, the more obvious the pain.

SECONDARY OUTCOMES:
The patient was followed up at 1 year after surgery to evaluate the International Hip Outcome Tool-12 (iHOT-12). | 1 year after operation
  The International Hip Outcome Tool-12 (iHOT-12).The highest score was 120, and the lowest was 0. The higher the score, the better the postoperative recovery.
The patient was followed up at 2 years after surgery to evaluate the International Hip Outcome Tool-12 (iHOT-12). | 2 years after operation
  The International Hip Outcome Tool-12 (iHOT-12).The highest score was 120, and the lowest was 0. The higher the score, the better the postoperative recovery.
The patient was followed up at 5 years after surgery to evaluate the International Hip Outcome Tool-12 (iHOT-12). | 5 years after operation
  The International Hip Outcome Tool-12 (iHOT-12).The highest score was 120, and the lowest was 0. The higher the score, the better the postoperative recovery.
The patient was followed up at 1 year after surgery to evaluate modified Harris Hip Score (mHHS). | 1 year after operation
  Modified Harris Hip Score (mHHS).The highest score was 44, and the lowest was 0. The higher the score, the better the postoperative recovery.
The patient was followed up at 2 years after surgery to evaluate modified Harris Hip Score (mHHS). | 2 years after operation
  Modified Harris Hip Score (mHHS).The highest score was 44, and the lowest was 0. The higher the score, the better the postoperative recovery.
The patient was followed up at 5 years after surgery to evaluate modified Harris Hip Score (mHHS). | 5 years after operation
  Modified Harris Hip Score (mHHS).The highest score was 44, and the lowest was 0. The higher the score, the better the postoperative recovery.

CONTACTS AND LOCATIONS:
Overall Officials: yan xu, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No